CLINICAL TRIAL: NCT02516072
Title: The Use of Remote Ischaemic Preconditioning in the Prevention of Contrast Induced Nephropathy in Patients Undergoing Elective Diagnostic or Therapeutic Peripheral Angiography: a Pilot Randomised Controlled Trial
Brief Title: Use of Remote Ischaemic Preconditioning in the Prevention of Contrast Induced Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: University College Hospital Galway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGH-RIPC
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Remote Ischaemic Preconditioning; Contrast Induced Nephropathy
Keywords: remote ischemic preconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients will receive iv hydration prior to procedure dependent on classification of risk as per eGFR.
- Remote Ischaemic preconditioning (RIPC) (Experimental): Patients will receive iv hydration prior to procedure dependent on classification of risk as per eGFR. Additionally, patients will receive RIPC; a blood pressure cuff will be placed around one arm of the patient, it will then be inflated to a pressure of 250mmHg for 5 minutes. The cuff will then be deflated and the arm allowed to reperfuse for 5 minutes. This will be repeated so that each patient receives a total of 3 ischaemia-reperfusion cycles immediately prior to the procedure.
  Interventions: Other: RIPC

INTERVENTIONS:
Other: RIPC — IV hydration prior to procedure dependent on classification of risk as per eGFR + RIPC
  Arms: Remote Ischaemic preconditioning (RIPC)

SUMMARY:
With an increasingly ageing population the incidence of peripheral arterial disease (PAD) is rising. With approximately one quarter of all PAD patients ultimately progressing to Critical Limb Ischaemia (CLI), increased demands are being placed on vascular imaging to accurately assess stenotic lesions. Early infrainguinal lesions (i.e. TASC A & B) can be treated with angioplasty+/- stenting and accurate assessment relies on the imaging gold standard of angiography.

Patients with PAD often have concomitant co morbidities such as diabetes and chronic renal impairment placing them at increased risk of developing contrast induced nephropathy (CIN) when exposed to iodinated contrast media. High risk individuals with decreased eGFR <60ml/min have a risk of between 20-30% of developing CIN. They have increased morbidity and mortality risks with a greater need for dialysis and prolonged in patient hospital stays. Ideally, the investigators should be searching for ways to decrease the incidence of CIN. Animal studies and more recently pilot human trials have shown that subjecting a remote vascular bed to a brief ischaemic stress, followed by a period of reperfusion; in what has been termed remote ischemic preconditioning (RIPC), may confer a protective benefit against the development of CIN. This study aims to determine if RIPC can protect against CIN in patients undergoing elective peripheral angiography for infrainguinal disease.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) affects between 3-10% of the population with prevalence rates rising with age to 15-20% in patients over 70 [1]. Worldwide incidence rates are rising, with the trend likely to persist with rising obesity and diabetes levels. Increasing numbers of affected patients require angiography as either a diagnostic or a therapeutic modality to improve peripheral blood flow and relieve the symptoms of CLI. The use of iodinated contrast medium during either diagnostic or therapeutic procedures can lead to contrast induced nephropathy (CIN) by direct toxic effects on renal tubular cells or by the induction of renal ischemia. Contrast induced nephropathy is a leading cause of hospital acquired acute kidney injury (AKI) and is defined as an acute deterioration in renal function as defined by the relative increase in serum creatinine levels >=25% or by a factor >=0.5mg/dl above baseline within 48 hours of administration of iv contrast in absence of other causes of renal dysfunction [2],[3]. While the incidence of CIN in the general population is only 2%, it rises in high risk patients to as high as 20-30% [4],[5]. Important risk factors for the development of CIN include pre-existing impaired renal function, diabetes mellitus, hypertension, increased age and congestive cardiac failure [5]. Depending on the risks present varying percentages of patients will proceed to require temporary or permanent dialysis, with inherently higher morbidity and mortality rates [5],[6],[7]. The identification and appropriate management of these patients to prevent CIN is important to decrease the associated accompanying morbidity and mortality in this patient cohort. Remote ischaemic preconditioning (RIPC) has been shown to confer benefit in both animal studies and in patients undergoing coronary angiography.

A large cohort study of 5787 patients with advanced PAD found that both moderate and severe renal insufficiency were associated with increased odds of death. The 1 year mortality risk was noted to be higher in patients with severe renal insufficiency (GFR<30ml/min per 1.73m2) (OR: 2.97 95%CI: 2.39-3.69) and they also tended to have a higher risk of presenting with tissue damage (ischemic ulceration or gangrene) compared with individuals having normal renal function (OR: 2.21; 95% CI: 0.64-2.98) [8].

Zaraca et al. in a recent systematic review reported on incidence of CIN of 9.2% in patients undergoing vascular surgery [9]. Identifiable risk factors included age >70yrs, high contrast volume, pre exisiting renal disease and the use of antihypertensive medication.

Ischaemic preconditioning is an endogenous mammalian mechanism whereby a brief period of ischaemia and reperfusion confers resistance to subsequent prolonged ischaemic insults. First observed in the canine heart, subsequent investigators noted that brief ischaemia in remote organs e.g. skeletal muscle induced protection in key central organs e.g. the heart. This remote ischaemic preconditioning (RIPC) does not require direct interference with the target organs' blood supply. It can be induced using blood pressure cuffs to produce brief episodes of upper limb ischaemia and reperfusion. It confers protection upon numerous organs simultaneously. RIPC reduces myocardial injury following aortic aneurysm repair, cardiac surgery and angioplasty. It also reduces adverse ischaemic events up to six months following percutaneous coronary intervention, implying some medium-term effect.

To date ischaemic conditioning has been applied primarily to the heart however animal studies have shown pre conditioning to offer renal protection [11],[12]. Although direct application of renal ischaemia is impractical, remote ischaemic conditioning applied prior to or during angiography procedures may offer protection to the kidneys against CIN. Whittaker and Przyklenk in 2011 explored this concept retrospectively using data from patients who had undergone emergency angioplasty for ST elevation myocardial infarction [13]. The original trial was a RCT which examined the protective effect of postconditioning on myocardial ischemia [14]. The authors retrospectively examined if study patients treated with multiple coronary balloon inflations had better renal function than patients not exposed to this remote conditioning. They concluded that patients in the conditioning group received 25% more contrast volume than the control group and showed no decline in renal function as demonstrated by examination of glomerular filtration rate at day 3 post procedure in comparison to the control group which saw a significant decline in renal function. Fikret et al in 2012 in the Renal Protection Trial demonstrated a protective benefit with RIPC from the development of CIN in high risk patients undergoing elective coronary angiography [15]. The need for contrast-based procedures is rising, especially in vascular surgery with increasing numbers of patients undergoing endovascular procedures, as is the incidence of post-contrast renal failure, which has a reported mortality of 34% [16]. The potential use of RIPC therefore to reduce the risk of kidney damage demands s further investigation in patients with advanced peripheral arterial disease who are at an increased risk of developing CIN.

ELIGIBILITY:
Inclusion Criteria:

* Elective intra-arterial peripheral angiography/angioplasty;
* Patients >21 years of age;
* Patients with CKD as evidenced by eGFR levels of 30ml/min < eGFR < 60ml/min (moderate risk) or eGFR levels of >= 60ml/min (low risk).

Exclusion Criteria:

* Severe renal impairment eGFR <30ml/min;
* Evidence of acute renal failure or patients on dialysis;
* History of previous CIN;
* Contraindication to volume replacement therapy;
* Pregnancy;
* Patients on glibenclamide or nicorandil (these medications may interfere with RIPC).

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12-30 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Reduction in the prevalence of contrast medium-induced nephropathy | At 24, 48 and 72 hours post procedure and 4-week post procedure
  Reduction is defined as an increase in the serum creatinine (serC) concentration of >25% from the baseline value within the 72-hour period after primary angiography.

SECONDARY OUTCOMES:
NGAL levels | At 2, 24, 48 and 72 hours post procedure
  mean NGAL level at 2-hour post procedure
Cystatin C levels | At 2, 24, 48 and 72 hours post procedure
  Mean changes of Cystatin C levels over 3 time points

OTHER OUTCOMES:
Length of hospital stay | 4 weeks post procedure
Need for dialysis | 4 weeks post procedure
  Free from dialysis
Mortality | 4 weeks post procedure
  Freedom from death

CONTACTS AND LOCATIONS:
Overall Officials: Tjun Yip Tang, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250